CLINICAL TRIAL: NCT00384839
Title: Phase II Study for the Use of Vidaza™ to Restore Responsiveness of Patients' Prostate Cancers to Hormonal Therapy
Brief Title: Vidaza to Restore Hormone Thx Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Celgene Corporation (Industry); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05015
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): azacitidine for injectable suspension
  Interventions: Drug: azacitidine for injectable suspension

INTERVENTIONS:
Drug: azacitidine for injectable suspension — Vidaza: 75 mg/m2 for 5 consecutive days (Days 1-5) of each 28 day cycle. A cycle will equal to 28 days. Patient will receive a maximum of 12 cycles.
  Other Names: Vidaza™

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) Vidaza has on patients with prostate cancer. This investigational drug is not approved by the Food and Drug Administration (FDA) for the treatment of prostate cancer; however, it is approved in myelodysplastic syndrome - a bone marrow disease. The pharmaceutical company involved in this study, Pharmion Corporation, is the manufacturer of Vidaza.

DETAILED DESCRIPTION:
This is an open label Phase II study. Patients will receive Vidaza for 5 consecutive days (Days 1- 5) of each 28-day cycle. Complete androgen ablation will be continued. Response will be assessed after a minimum of 2 cycles (evaluable patients). PSA response will be evaluated prior to each cycle and % fetal hemoglobin will be evaluated prior to each odd cycle (excluding Cycle 1). Patients will be treated until clinical progression up to a maximum of 12 cycles. A total of 35 patients with advanced metastatic HRPC will be enrolled in this trial.

ELIGIBILITY:
INCLUSION CRITERIA:

* A diagnosis of histologically confirmed, progressive, advanced metastatic, or nonmetastatic prostate cancer with documented PSA progression, with a calculated PSA doubling time <3 months, on complete androgen ablation therapy. PSA progression, with or without clinical progression (symptomatic/radiologic as per RECIST) is required; measurable disease is not required.

Baseline PSA values must be followed by 2 serial increases at least 2 weeks apart (no upper limit for time for these 2 samples). Calculated PSA doubling time, for the above PSA values must be <3 months. An automated PSA doubling time calculator may be found at www.mskcc.org/mskcc/html/10088.cfm (see study tools).

* Currently on complete androgen ablation hormone therapy (an LHRH agonist plus an antiandrogen) with testosterone level <50ng/dL). Patients who are on LHRH agonist or other antiandrogenic therapy at entry will continue that therapy while on this study. Anti-androgen withdrawal is not necessary and is precluded before enrollment on the trial. The details of that therapy must be recorded in the CRF. Patients who have had an orchiectomy and who are on antiandrogen therapy are permitted on study.
* An elevated PSA level for patients progressing by PSA criteria is required (see protocol for specific detail).
* Has a Karnofsky Performance Status >70
* Is greater than 18 years of age
* Must meet specific lab values for the following criteria: granulocyte, platelet count, total bilirubin, AST and ALT, serum creatinine, calculated creatinine clearance & urinalysis (see protocol for specific detail).
* If fertile, the patient has agreed to use an acceptable method of birth control to avoid fathering a child for the duration of the study and for a period of 2 months thereafter.
* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form

EXCLUSION CRITERIA:

* Has only clinical progression without evidence of PSA progression
* Has received prior chemotherapy
* Has had prior treatment with Vidaza
* Has a history of hypersensitivity to any component of Vidaza (mannitol)
* Has a history of New York Heart Association (NYHA) heart disease Class III or IV (Appendix III) or myocardial infarction within 6 months prior to Day 1 or unstable arrhythmia or evidence of ischemia on electrocardiogram (ECG)
* Is receiving concurrent immunotherapy
* Is receiving concurrent bisphosphonate therapy; long-standing bisphosphonate therapy (initiated >8 weeks prior to registration) is acceptable. Bisphosphonates started within the prior 8 weeks will not be allowed since this may affect other study endpoints and render their interpretation difficult.
* Has received treatment with radiation therapy, surgery, chemotherapy, ketoconazole, corticosteroids, or an investigational agent within 1 month prior to registration, (6 weeks for radiation therapy, nitrosureas or Mitomycin C)
* Has evidence of central nervous system (CNS) involvement
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection that requires systemic therapy
* Has a serious uncontrolled nonmalignant disease (liver failure, or other condition) that could compromise protocol objectives in the opinion of the Investigator
* Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin), which could affect the diagnosis or assessment of any of the study drugs
* Is known to be positive for the human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Is unable to comply with requirements of study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guru Sonpavde, MD, Principal Investigator — US Oncology Research
Locations (13):
- United States (13):
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - Raleigh Hematology Oncology Associates, Cary, North Carolina
  - Northwestern Carolina Oncology Hematology, Hickory, North Carolina
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Cancer Care Nrothwest-South, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Vidaza: azacitidine for injectable suspension : Vidaza: 75 mg/m2 for 5 consecutive days (Days 1-5) of each 28 day cycle. A cycle will equal to 28 days. Patient will receive a maximum of 12 cycles.
Period: Overall Study
Arm/Group | Vidaza
Started | 36
Completed | 28
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Investigator Request | 1
Not completed — Patient Request | 1
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Population: ITT Population
Arm/Group | Vidaza
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 33
  Hispanic | 2
  Black | 1
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With PSA Doubling Time >=3 Months.
Description: To determine if Vidaza can convert hormone-refractory prostate cancer to a hormone-responsive state. This will be assessed by the proportion of patients who have a documented prostate specific antigen (PSA) doubling time >3= months.
Time Frame: Until progression or up to a maximum of 12 cycles
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: % of patients with PSA-DT>= 3 months
Arm/Group | Vidaza
Number analyzed (Participants) | 34
% of patients with PSA-DT>= 3 months | 55.8 [37.9 to 72.8]

2. Secondary Outcome: PSA Response Rate
Description: Complete PSA Response defined as complete normalization of PSA maintained for at least 4 weeks, and partial PSA response defined as a decrease in PSA level of at least 50% from baseline level maintained for at least 4 weeks.
Time Frame: Every 8 weeks for 1 year.
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vidaza
Number analyzed (Participants) | 34
percentage of participants | 0 [0 to 0]

3. Secondary Outcome: Objective Response Rate by Recist (ORR)
Description: ORR = Complete Response (CR) + Parcial response (PR). CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: Every 8 weeks for 1 year.
Population: Only for patients with lesions evaluable by RECIST criteria at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vidaza
Number analyzed (Participants) | 13
percentage of participants | 0 [0 to 0]

4. Secondary Outcome: Progression-free Survival
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 1.5 year.
Population: ITT population
Measure: Median (Full Range); unit: weeks
Arm/Group | Vidaza
Number analyzed (Participants) | 36
weeks | 12.4 [2.1 to 70.3]

5. Secondary Outcome: 1-year Overall Survival (OS)
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: Up to 1 year.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Probability of Survival at 1-year
Arm/Group | Vidaza
Number analyzed (Participants) | 36
Probability of Survival at 1-year | 0.73 [0.54 to 0.85]

6. Secondary Outcome: Changes in Fetal Hemoglobin (HbF) With Time.
Description: Time from baseline to maximal fetal hemoglobin (HbF).
Time Frame: Up to 1 year.
Population: Patients with HbF measurements.
Measure: Median (Full Range); unit: weeks
Arm/Group | Vidaza
Number analyzed (Participants) | 14
weeks | 12.7 [8.4 to 26.6]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | Vidaza
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 31/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vidaza (N=34)
NAUSEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vidaza (N=34)
ANEMIA (Blood and lymphatic system disorders) | 7 (9)
ANOREXIA (Gastrointestinal disorders) | 7 (7)
CONSTIPATION (Gastrointestinal disorders) | 13 (16)
CREATININE SERUM INCREASED (Metabolism and nutrition disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 3 (3)
FATIGUE (General disorders) | 14 (16)
INJECTION SITE PAIN (Skin and subcutaneous tissue disorders) | 2 (4)
INJECTION SITE REACTION (Skin and subcutaneous tissue disorders) | 9 (19)
LEUCOPENIA (Blood and lymphatic system disorders) | 3 (11)
NAUSEA (Gastrointestinal disorders) | 11 (14)
NEUROPATHY (Nervous system disorders) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 6 (11)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 3 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (3)
VOMITING (Gastrointestinal disorders) | 10 (11)
WEAKNESS (General disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Further development of azacitidine in patients with prostate cancer may be warranted in randomized trials, alone and in combination with hormonal therapy, chemotherapy and histone deacytelase inhibitors

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No